CLINICAL TRIAL: NCT06953505
Title: Pilot Study of At Home Ammonia Monitoring in Patients With an Inborn Error of Ammonia Metabolism
Brief Title: At Home Ammonia Monitoring of Inborn Errors of Ammonia Metabolism
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sequitur Health Corp. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HD112243; 1R44HD112243 (NIH); STUDY00025898 (Other: Oregon Health & Science University)
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Urea Cycle Disorders; Organic Acidemias; Fatty Acid Oxidation Disorder; Ammonia; Metabolic Disorder
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Ammonia Device (Experimental)
  Interventions: Diagnostic Test: Ammonia Study Device

INTERVENTIONS:
Diagnostic Test: Ammonia Study Device — Ammonia study device for capillary ammonia measurement

SUMMARY:
The goal of this observational study is to learn if people with certain ammonia metabolism disorders will measure their ammonia levels at home.

The main question it aims to answer is:

• Will participants measure their ammonia every day?

Participants will be asked to:

* Attend three in-person study visits at the clinic.
* Measure temperature, heart rate, and blood oxygen every day.
* Complete a short survey every day.
* Measure ammonia every day.

DETAILED DESCRIPTION:
Ammonium (NH4+, ion in aqueous solution) exists in equilibrium with ammonia (NH3, gas) according to the equilibrium reaction: NH3+ + H+ ↔ NH4+, which has a pKa of 9.25.[1] Total ammonia is the sum of all ammonium ions (NH4+) and ammonia gas (NH3) present. At the physiologically relevant pH of blood (~7.4), the ammonium/ammonia equilibrium is almost completely shifted to NH4+.[2] Total ammonia is colloquially referred to as ammonia in clinical medicine and clinical chemistry. Thus, the term ammonia in this document refers to total ammonia unless otherwise specified.

Ongoing metabolic processes in the human body continuously generate ammonia.[1,3-8] Ammonia is produced in all tissues of the body, mainly by the process of transamination followed by deamination, from biogenic amines and amino groups of nitrogenous bases (e.g., purines, pyrimidines), and within the intestine by intestinal bacterial flora through the action of urease on urea.[1, 7] Much of the ammonia produced in the intestine travels to the liver via the portal circulation. Ammonia produced by the kidneys variably clears the body in urine or enters the systemic circulation via the renal veins.[7-9]

Ammonia levels within an individual are highly dynamic over the course of a day based on dietary and exercise status.

Because of the dynamic ongoing metabolic cellular processes that generate and dispose of ammonia, accurate measurement of ammonia can be challenging; cellular components in blood may continue to create ammonia after the blood is drawn, amino acids may deaminate nonenzymatically or enzymatically. Blood samples should be immediately measured. If not immediately measured, then blood samples should be kept on ice and measured within 30 minutes of collection.

Ammonia is toxic to the central nervous system.[10]

Increased ammonia within the blood (hyperammonemia) may be caused by a variety of factors, including:

Conditions associated with either acute or chronic liver dysfunction, including, but not limited to:

Non-viral hepatitis (e.g., autoimmune hepatitis, alcoholic hepatitis, drug-induced hepatitis, ischemic hepatitis) Viral hepatitis (e.g., A, B, C, D, E, cytomegalovirus (CMV), Epstein-Barr virus (EBV) rubella (measles)) Reye's syndrome Cirrhosis End Stage Liver Disease

Certain inborn errors of metabolism including, but not limited to:

Urea cycle disorders Organic acidemias Fatty acid oxidation disorders Gastrointestinal bleeding Certain infections (including those caused by urease-producing bacteria)

Various medications, including, but not limited to:

Valproic acid Topiramate Carbamazepine Measurable changes in cognition may be associated with hyperammonemia. With either acute or chronic liver dysfunction, hepatic encephalopathy or hepatic coma may occur with hyperammonemia.

With an inborn error of metabolism affecting ammonia metabolism, a hyperammonemic crisis may occur with hyperammonemia.

Ammonia levels may increase with increasing dietary protein intake. Ammonia levels can vary throughout the day.

This Ammonia Device consists of a reusable instrument and a single-use cartridge based system that accepts a single drop of whole blood. It operates on the photometric method. The System measures the color change of a dye in the Cartridge in response to the amount of ammonia in a fixed volume of sample. Ammonia Device system. This is an investigational use only device and the performance characteristics of this product have not been established.

[ 1 ] Adeva, M. M.; Souto, G.; Blanco, N.; Donapetry, C. Ammonium metabolism in humans. Metabolism 2012, 61 (11), 1495-1511. DOI: 10.1016/j.metabol.2012.07.007.

[ 2 ] Bates, R. G.; Pinching, G. D. Acidic Dissociation Constant of Ammonium Ion at 0 to 50°C and the Base Strength of Ammonia. Journal of Research of the National Bureau of Standards 1949, 42, 419-430. DOI: 10.6028/jres.042.037.

[ 3 ] Patel, R.; Kaemingk, B. D.; Carey, W. A.; Block, D. R.; Madigan, T. Proposed Plasma Ammonia Reference Intervals in a Reference Group of Hospitalized Term and Preterm Neonates. The Journal of Applied Laboratory Medicine 2020, 5 (2), 363-369. DOI: 10.1093/jalm/jfz001.

[ 4 ] Berry, S. A.; Lichter-Konecki, U.; Diaz, G. A.; McCandless, S. E.; Rhead, W.; Smith, W.; LeMons, C.; Nagamani, S. C. S.; Coakley, D. F.; Mokhtarani, M.; et al. Glycerol phenylbutyrate treatment in children with urea cycle disorders: Pooled analysis of short and long-term ammonia control and outcomes. Molecular Genetics and Metabolism 2014, 112 (1), 17-24. DOI: 10.1016/j.ymgme.2014.02.007.

[ 5 ] Häberle, J.; Burlina, A.; Chakrapani, A.; Dixon, M.; Karall, D.; Lindner, M.; Mandel, H.; Martinelli, D.; Pintos-Morell, G.; Santer, R.; et al. Suggested guidelines for the diagnosis and management of urea cycle disorders: First revision. Journal of Inherited Metabolic Disease 2019, 42 (6), 1192-1230. DOI: 10.1002/jimd.12100.

[ 6 ] Lee, B.; Diaz, G. A.; Rhead, W.; Lichter-Konecki, U.; Feigenbaum, A.; Berry, S. A.; Le Mons, C.; Bartley, J. A.; Longo, N.; Nagamani, S. C.; et al. Blood ammonia and glutamine as predictors of hyperammonemic crises in patients with urea cycle disorder. Genet Med 2015, 17 (7), 561-568. DOI: 10.1038/gim.2014.148 From NLM.

[ 7 ] Weiner, I. D.; Hamm, L. L. Molecular mechanisms of renal ammonia transport. Annu Rev Physiol 2007, 69, 317-340. DOI: 10.1146/annurev.physiol.69.040705.142215.

[ 8 ] Levitt, D. G.; Levitt, M. D. A model of blood-ammonia homeostasis based on a quantitative analysis of nitrogen metabolism in the multiple organs involved in the production, catabolism, and excretion of ammonia in humans. Clin Exp Gastroenterol 2018, 11, 193-215. DOI: 10.2147/CEG.S160921.

[ 9 ] Mohiuddin, S. S.; Khattar, D. Biochemistry, Ammonia. In StatPearls, 2025. [ 10 ] Balistreri, W.; Rej, R. Liver Function. In Tietz Fundamentals of Clinical Chemistry. 4th ed.Philadelphia, Burtis, C., Ashwood, E. Eds.; WB Saunders, 1996; pp 539-568.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed ammonia disorder such as

  * Ornithine transcarbamylase deficiency
  * Systemic primary carnitine deficiency
  * Type I citrullinemia
  * Argininosuccinic aciduria
  * Isolated methylmalonic acidemia
  * Type II citrullinemia
  * Propionic acidemia
  * Isovaleric acidemia
  * Multiple acyl-CoA dehydrogenase deficiency
  * Pyruvate carboxylase deficiency
  * Argininemia (arginase deficiency)
  * Carbamoyl phosphate synthase I deficiency
  * Dihydrolipoamide dehydrogenase deficiency
  * Lysinuric protein intolerance
  * Hyperornithinemia-hyperammonemia-homocitrullinuria
  * Carnitine-acylcarnitine translocase deficiency
  * Carbonic anhydrase VA deficiency
  * N-acetyl glutamate synthetase deficiency
* English Literacy

Exclusion Criteria:

* Incarcerated
* Presence of a non-inborn error of metabolism medical condition associated with abnormal ammonia metabolism (e.g., end stage liver disease).
* Unable to read in English

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of daily ammonia measurements completed. | through individual participant study completion - approximately 240 days per participant with an optional 120 day additional extension period available.
  Daily ammonia measurements will be completed on the ammonia study device. A single participant will have a single device. The device will store information about the time, date, and results from the measurements completed. The primary hypothesis is that participants will complete 90% of the daily ammonia measurements during their individual study periods.

SECONDARY OUTCOMES:
Descriptive Statistics and Correlations | From enrollment through study completion, this is an average of 240 days per participant. If a participant chooses to participate in the optional study extension then the time frame will be approximately 360 days per participant.
  After the study is complete, descriptive statistics (mean, median, range) will be calculated for individual participants for the study for the quantitative home measurements (temperature, heart rate, pulse oxygenation, and capillary ammonia). Descriptive statistics (mean, median, range) will be calculated for all aggregated participant data for the study for the quantitative home measurements (temperature, heart rate, pulse oxygenation, and capillary ammonia). The strength of correlations between quantitative values and participant self reported survey information and/or medical record documented clinical events will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Marylaura L Thomas, Ph.D., Principal Investigator — Sequitur Health Corp.; Leslie F. Thomas, M.D., Study Director — Sequitur Health Corp.
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified primary outcome participant data sets for results used in publications will be made available for sharing at the time the results are published in a peer-review publication.
  Deidentified secondary outcome participant data sets will be made available upon request to Sequitur Health Corp. after a data sharing agreement is signed.
Supporting Information: Study Protocol, ICF
Time Frame: Upon publication in a peer-reviewed publication and in perpetuity once the publication is available.
Access Criteria: All peer reviewed publications will be published open-access so anyone with an internet connection will be able to access the publication, the data contained within the publication, and any supplementary information to the publication.
  Secondary outcome individual participant data that may not be included in a publication will be made available after a data sharing agreement is executed between the receiving party and Sequitur Health Corp.. To request secondary outcome data, after the completion of the study, please contact Sequitur Health Corp. at info@sequiturhealth.com or 1-855-445-3889.

DOCUMENTS (4):
  • Informed Consent Form: Child Assent Form (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT06953505/ICF_001.pdf
  • Informed Consent Form: Adult Consent Form (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT06953505/ICF_000.pdf
  • Informed Consent Form: Adult Consent Form - revised 9/23/2025 (2025-09-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT06953505/ICF_002.pdf
  • Informed Consent Form: Child Assent Form - revised 9/23/2025 (2025-09-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT06953505/ICF_003.pdf